CLINICAL TRIAL: NCT06494007
Title: Reducing Diltiazem-Related Hypotension in Atrial Fibrillation: The Role of IV Calcium Pretreatment
Brief Title: Role of IV Calcium to Prevent Diltiazem-related Hypotension
Acronym: AFstd
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Adem Az, Medical Doctor, Haseki Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Haseki TRH
Record Dates: First submitted 2024-07-01; First posted 2024-07-10 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation; Rapid Ventricular Response; Hypotension Drug-Induced
Keywords: Atrial fibrillation; Rapid ventricular response; Diltiazem-related hypotension; IV Calcium
MeSH Terms: conditions — Atrial Fibrillation; Hypotension | interventions — Sodium Chloride; Calcium

STUDY DESIGN:
Intervention Model Description: Single center
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Each participant was assigned an identification number indicating their treatment group. An emergency nurse prepared the treatment solutions just before administration based on the assigned identification number and stored them in labeled containers with no indication of their content. A clinician with eight years of experience, who was blinded to the study's null hypothesis and did not participate in the evaluation of results, administered the treatments and recorded patient data onto a pre-prepared case data form. Another physician, who was not present during the treatment, assessed the findings post-treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Diltiazem monotherapy (Active Comparator): The Diltiazem monotherapy
  Interventions: Drug: Sodium chloride
- Diltiazem with 90 mg calcium (Active Comparator): Diltiazem with 90 mg calcium
  Interventions: Drug: 90 mg of calcium
- The Diltiazem with 180 mg calcium (Active Comparator): Diltiazem with 180 mg calcium
  Interventions: Drug: 180 mg Calcium

INTERVENTIONS:
Drug: Sodium chloride — The Diltiazem monotherapy group received 6.66 mL of IV sodium chloride 0.9% (NaCl) prior to receiving IV weight-adjusted diltiazem.
  Arms: Diltiazem monotherapy
Drug: 90 mg of calcium — The Diltiazem with 90 mg calcium group received 3.33 mL of IV calcium chloride (CaCl2, 90 mg) and 3.33 mL of IV NaCl 0.9% as pretreatment over 5-10 min prior to receiving IV diltiazem.
  Arms: Diltiazem with 90 mg calcium
Drug: 180 mg Calcium — The Diltiazem with 180 mg calcium group received 6.66 mL of IV CaCl2 (180 mg) as pretreatment prior to receiving IV diltiazem.
  Arms: The Diltiazem with 180 mg calcium

SUMMARY:
The objective of this study is to examine the efficacy and safety of IV calcium pretreatment at varying doses prior to weight-adjusted IV Diltiazem on the incidence of Diltiazem-related hypotension in adult patients presenting to the Emergency Department due to Atrial Fibrillation with Rapid Ventricular Response. Specifically, we tested the hypothesis that patients with Atrial Fibrillation who receive IV calcium pretreatment prior to IV Diltiazem suffer less hypotension than those receiving Diltiazem monotherapy.

DETAILED DESCRIPTION:
Patients were randomly divided into one of three groups. We assessed the Systolic Blood Pressure and Heart Rate of participants before treatment and 5, 10, and 15 min after treatment among the patient groups. Successful rhythm control was defined as achieving an HR of <100 bpm, a reduction in HR by >20% compared to baseline, or the restoration of normal sinus rhythm (NSR). If adequate rhythm control was not achieved within 15 min of the initial treatment, we administered 0.35 mg/kg of IV diltiazem slowly over 2 minutes as a rescue treatment. The need for rescue treatment or any intervention for hypotension, as well as any adverse effects, were recorded in a prepared data form. Also, patient demographics (age and sex), new onset versus chronic AFib/AFL, relevant medical history, vital signs on admission (SBP and HR), complaints and symptoms on admission, and laboratory parameters were documented in a prepared data form.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients with documented AFib/AFL (confirmed by ECG)
* Patients with a Heart Rate of ≥ 120 bpm, and a Systolic Blood Pressure of ≥ 90 mmHg

Exclusion Criteria:

* Patients under 18 years of age
* pregnant individuals
* Patients with hemodynamic instability requiring electrocardioversion
* Patients with a documented history of sick sinus syndrome, third-degree AV block, Wolff-Parkinson-White syndrome
* Patients with hypotension (SBP <90 mmHg)
* Patients with known or suspected hypercalcemia
* Patients with a confirmed allergy to diltiazem
* Patients with concurrent use of another Heart Rate control agent (such as beta-blockers, amiodarone, or digoxin) on the same admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Change in Systolic blood pressure before and after treatment | 5, 10, and 15 minutes following the initial administration.
  We investigated the change in systolic blood pressure at 5, 10, and 15 minutes following the initial IV diltiazem administration comparatively among treatment groups.

SECONDARY OUTCOMES:
Change in Heart Rate before and after treatment | 5, 10, and 15 minutes following the initial administration
  We also investigated the change in Heart rate values at 5, 10, and 15 minutes following the initial IV diltiazem administration comparatively among treatment groups.

OTHER OUTCOMES:
Assessing the treatment-related complications | 2 hours following the initial administration
  We also evaluated treatment-related adverse effects, hypotension, and hypercalcemia.

CONTACTS AND LOCATIONS:
Overall Officials: Adem Az, M.D., Principal Investigator — Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Stored in non-publicly available Available on request

REFERENCES:
- [Result] Rossi N, Allen B, Hailu K, Kamataris K, Ryan C. Impact of intravenous calcium with diltiazem for atrial fibrillation/flutter in the emergency department. Am J Emerg Med. 2023 Feb;64:57-61. doi: 10.1016/j.ajem.2022.11.018. Epub 2022 Nov 17. PMID 36442264
- [Result] Kolkebeck T, Abbrescia K, Pfaff J, Glynn T, Ward JA. Calcium chloride before i.v. diltiazem in the management of atrial fibrillation. J Emerg Med. 2004 May;26(4):395-400. doi: 10.1016/j.jemermed.2003.12.020. PMID 15093843
- [Result] Jameson SJ, Hargarten SW. Calcium pretreatment to prevent verapamil-induced hypotension in patients with SVT. Ann Emerg Med. 1992 Jan;21(1):68. doi: 10.1016/s0196-0644(05)82242-5. No abstract available. PMID 1539892
- [Result] Lipman J, Jardine I, Roos C, Dreosti L. Intravenous Calcium chloride as an antidote to verapamil-induced hypotension. Intensive Care Med. 1982 Jan;8(1):55-7. doi: 10.1007/BF01686855. No abstract available. PMID 7056937
- [Derived] Az A, Sogut O, Dogan Y, Akdemir T, Ergenc H, Umit TB, Celik AF, Armagan BN, Bilici E, Cakmak S. Reducing diltiazem-related hypotension in atrial fibrillation: Role of pretreatment intravenous calcium. Am J Emerg Med. 2025 Feb;88:23-28. doi: 10.1016/j.ajem.2024.11.033. Epub 2024 Nov 17. PMID 39577214